CLINICAL TRIAL: NCT01138462
Title: Universal Screening and Decolonization vs Standard Precautions for Control of Methicillin-resistant Staphylococcus Aureus (MRSA) in Nursing Homes: a Cluster, Randomised Controlled Study.
Brief Title: Control of MRSA in Nursing Homes: Decolonization vs Standard Precautions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Bellini Cristina, MD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocole 96/10
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: Methicillin-Resistant Staphylococcus aureus; Decolonisation; Nursing homes; Infection Control
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Precautions (No Intervention): control arm, standards precautions for all residents living in the nursing home of control arm, including MRSA carriers
- Intervention (Other): Intervention arm, standards precautions for all residents living in nursing homes of intervention arm, and topical decolonization for MRSA carriers, including environmental disinfection
  Interventions: Other: intervention

INTERVENTIONS:
Other: intervention — 5 days topical decolonisation including nasal mupirocin tid, chlorhexidine mouth wash tid, chlorhexidine body wash once daily.
  Daily direct resident's environmental disinfection during decolonisation.
  Other Names: topical MRSA decolonisation and environmental disinfection
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the better approach between the currently procedure (i.e. standards precautions) and a reinforced strategy to control MRSA transmission in the institutionalized population of nursing homes in Canton of Vaud, Switzerland.

DETAILED DESCRIPTION:
MRSA carriage among nursing homes residents of Canton Vaud, Switzerland, is increasing, despite use of standard precautions. Recommendation to prevent MRSA transmission in long term care facilities are lacking. We aim to reinforce the current infection control strategy by general MRSA screening of institutionalised residents and decolonisation of MRSA carriers. Because the uncertainties in the impact of this reinforced strategy, we aim to compare this action to the policy actually applied.

ELIGIBILITY:
Inclusion Criteria:

* all nursing homes of canton Vaud, Switzerland, that give the consent of participation

Exclusion Criteria:

- refusal to participate

Inclusion criteria for decolonisation in intervention nursing homes:

- all MRSA positive residents living in a Nursing Home included in the intervention group

Exclusion Criteria for decolonisation:

* residents that refuse to be screened or refused the decolonisation
* life expectancy shorter of 7 days
* known intolerance of disinfectant/ topical antibiotics used in the protocol
* active MRSA infection
* asymptomatic MRSA bacteriuria
* stage IV wound (according to National Pressure Ulcer Advisory Panel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the change in prevalence of MRSA carriage among residents of each Nursing homes group at the end of the one study year | 1 year
  in each control and intervention nursing home: MRSA screening of all residents of nursing homes of Canton Vaud, at baseline and 1 year later, in order to compare MRSA prevalence changes at nursing homes levels

SECONDARY OUTCOMES:
To determine the effectiveness of the reinforced strategy to prevent MRSA infection, compared to the standard strategy | 1 year
  In a subpopulation of all nursing homes residents (10% of the whole population), recording of all microbiologically documented MRSA infection, according to nosocomial infection definitions of the Center of Diseases Control (CDC) of Atlanta.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Zanetti, MD, Study Director — University Hospital of Lausanne, Switzerland

REFERENCES:
- [Background] Bellini C, Petignat C, Masserey E, Bula C, Burnand B, Rousson V, Blanc DS, Zanetti G. Universal screening and decolonization for control of MRSA in nursing homes: a cluster randomized controlled study. Infect Control Hosp Epidemiol. 2015 Apr;36(4):401-8. doi: 10.1017/ice.2014.74. PMID 25782894